CLINICAL TRIAL: NCT00594477
Title: Intensity Modulated Radiation Therapy for Breast Cancer: A Phase I Feasibility Study
Brief Title: Intensity Modulated Radiotherapy for Breast Cancer
Acronym: IMRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-1077 / 201106403
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: IMRT; breast cancer with regional nodal metastasis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IMRT (Experimental): The prescribed dose for all patients will be 5040 cGy in 28 fractions. Patients will receive external beam treatment once a day, five days a week for approximately five and a half weeks.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT

SUMMARY:
This study delivers radiation therapy to any residual breast tissue and the chest wall plus lymph node areas around the breast. These lymph node areas are under the arm, around the collar bone, and under the sternum (breastbone).

DETAILED DESCRIPTION:
IMRT treatment uses a computer-controlled x-ray (CT) to deliver radiation beams at several different angles and strengths to deliver precise doses to the regions at risk for recurrence of breast cancer while reducing or sparing the dose to critical structures (heart, lungs) and nearby normal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥ 18 years
* Invasive primary female breast cancer
* Pathologically proven regional nodal metastasis
* Status post mastectomy or partial mastectomy with an assessment of axillary nodes via sentinel lymph node biopsy and/or axillary lymph node dissection.
* Signed study specific consent form

Exclusion Criteria:

* Distant metastasis
* Currently Pregnant
* Psychiatric or addictive disorders that preclude informed consent
* Time from initial diagnosis to the start of radiation therapy > one year
* Estimated life expectancy judged to be < one year
* Prior radiation to the ipsilateral breast or chest wall
* Primary breast cancer is lymphoma or sarcoma
* Patients being treated with concurrent chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-01-04 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of adjuvant comprehensive radiation therapy via IMRT with daily set-up position verified using 3D verification | Within 1 year of protocol registration
  The study will be deemed infeasible if greater than 10% of enrolled patients have at least one of the following outcomes:
  1. Patient cannot be given the treatment because her anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised for her.
  2. Within 1 year of protocol registration, the patient develops radiation pneumonitis toxicity of greater than or equal to grade 3 by CTCAE scales.
  3. Within 1 year of protocol registration, the patient develops any local or regional breast cancer recurrence.
  4. Within 1 year of protocol registration, the patient dies from causes judged to be related to her treatment.

SECONDARY OUTCOMES:
Evaluate the rate and severity of both acute and late cutaneous toxicity | 6-8 months following completion of treatment and 12-14 months following completion of treatment
Evaluate the rate and severity of late subcutaneous fibrosis | 6-8 months following completion of treatment and 12-14 months following completion of treatment
Evaluate the rate of radiation pneumonitis | 6-8 weeks following completion of treatment, 3-4 months following completion of treatment, 6-8 months following completion of treatment, and 12-14 months following completion of treatment
Evaluate ipsilateral upper quadrant function | Pretreatment and 3-4 months following completion of treatment
  For patients who receive physical therapy, objective measures of the rotator cuff, bursa, and joint space will be evaluated by diagnostic ultrasound if medically indicated.
Evaluate patient quality of life | Pretreatment, 6-8 months following completion of treatment, and 12-14 months following completion of treatment
Evaluate local-regional control rates | 12-14 months following completion of radiation therapy
Evaluate patient set-up reproducibility in breast cancer patients treated with IMRT using daily 3D position verification | 12-14 months following completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Imran Zoberi, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El Moussaoui R, Opmeer BC, Bossuyt PM, Speelman P, de Borgie CA, Prins JM. Development and validation of a short questionnaire in community acquired pneumonia. Thorax. 2004 Jul;59(7):591-5. doi: 10.1136/thx.2003.015107. PMID 15223867
- [Background] Ragaz J, Jackson SM, Le N, Plenderleith IH, Spinelli JJ, Basco VE, Wilson KS, Knowling MA, Coppin CM, Paradis M, Coldman AJ, Olivotto IA. Adjuvant radiotherapy and chemotherapy in node-positive premenopausal women with breast cancer. N Engl J Med. 1997 Oct 2;337(14):956-62. doi: 10.1056/NEJM199710023371402. PMID 9309100
- [Background] Ragaz J, Olivotto IA, Spinelli JJ, Phillips N, Jackson SM, Wilson KS, Knowling MA, Coppin CM, Weir L, Gelmon K, Le N, Durand R, Coldman AJ, Manji M. Locoregional radiation therapy in patients with high-risk breast cancer receiving adjuvant chemotherapy: 20-year results of the British Columbia randomized trial. J Natl Cancer Inst. 2005 Jan 19;97(2):116-26. doi: 10.1093/jnci/djh297. PMID 15657341
- [Background] Overgaard M, Hansen PS, Overgaard J, Rose C, Andersson M, Bach F, Kjaer M, Gadeberg CC, Mouridsen HT, Jensen MB, Zedeler K. Postoperative radiotherapy in high-risk premenopausal women with breast cancer who receive adjuvant chemotherapy. Danish Breast Cancer Cooperative Group 82b Trial. N Engl J Med. 1997 Oct 2;337(14):949-55. doi: 10.1056/NEJM199710023371401. PMID 9395428
- [Background] Overgaard M, Jensen MB, Overgaard J, Hansen PS, Rose C, Andersson M, Kamby C, Kjaer M, Gadeberg CC, Rasmussen BB, Blichert-Toft M, Mouridsen HT. Postoperative radiotherapy in high-risk postmenopausal breast-cancer patients given adjuvant tamoxifen: Danish Breast Cancer Cooperative Group DBCG 82c randomised trial. Lancet. 1999 May 15;353(9165):1641-8. doi: 10.1016/S0140-6736(98)09201-0. PMID 10335782
- [Background] Clarke M, Collins R, Darby S, Davies C, Elphinstone P, Evans V, Godwin J, Gray R, Hicks C, James S, MacKinnon E, McGale P, McHugh T, Peto R, Taylor C, Wang Y; Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of radiotherapy and of differences in the extent of surgery for early breast cancer on local recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 Dec 17;366(9503):2087-106. doi: 10.1016/S0140-6736(05)67887-7. PMID 16360786
- [Background] Fowble B, Gray R, Gilchrist K, Goodman RL, Taylor S, Tormey DC. Identification of a subgroup of patients with breast cancer and histologically positive axillary nodes receiving adjuvant chemotherapy who may benefit from postoperative radiotherapy. J Clin Oncol. 1988 Jul;6(7):1107-17. doi: 10.1200/JCO.1988.6.7.1107. PMID 3292711
- [Background] Truong PT, Woodward WA, Buchholz TA. Optimizing locoregional control and survival for women with breast cancer: a review of current developments in postmastectomy radiotherapy. Expert Rev Anticancer Ther. 2006 Feb;6(2):205-16. doi: 10.1586/14737140.6.2.205. PMID 16445373
- [Background] Huang EH, Strom EA, Perkins GH, Oh JL, Chen AM, Meric-Bernstam F, Hunt KK, Sahin AA, Hortobagyi GN, Buchholz TA. Comparison of risk of local-regional recurrence after mastectomy or breast conservation therapy for patients treated with neoadjuvant chemotherapy and radiation stratified according to a prognostic index score. Int J Radiat Oncol Biol Phys. 2006 Oct 1;66(2):352-7. doi: 10.1016/j.ijrobp.2006.04.046. Epub 2006 Aug 2. PMID 16887286
- [Background] Huang EH, Tucker SL, Strom EA, McNeese MD, Kuerer HM, Hortobagyi GN, Buzdar AU, Valero V, Perkins GH, Schechter NR, Hunt KK, Sahin AA, Buchholz TA. Predictors of locoregional recurrence in patients with locally advanced breast cancer treated with neoadjuvant chemotherapy, mastectomy, and radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):351-7. doi: 10.1016/j.ijrobp.2004.09.056. PMID 15890574
- [Background] Pierce LJ, Butler JB, Martel MK, Normolle DP, Koelling T, Marsh RB, Lichter AS, Fraass BA. Postmastectomy radiotherapy of the chest wall: dosimetric comparison of common techniques. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1220-30. doi: 10.1016/s0360-3016(01)02760-2. PMID 11955732
- [Background] Shapiro CL, Recht A. Side effects of adjuvant treatment of breast cancer. N Engl J Med. 2001 Jun 28;344(26):1997-2008. doi: 10.1056/NEJM200106283442607. No abstract available. PMID 11430330
- [Background] Favourable and unfavourable effects on long-term survival of radiotherapy for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 2000 May 20;355(9217):1757-70. PMID 10832826
- [Background] Paszat LF, Mackillop WJ, Groome PA, Boyd C, Schulze K, Holowaty E. Mortality from myocardial infarction after adjuvant radiotherapy for breast cancer in the surveillance, epidemiology, and end-results cancer registries. J Clin Oncol. 1998 Aug;16(8):2625-31. doi: 10.1200/JCO.1998.16.8.2625. PMID 9704712
- [Background] Hojris I, Overgaard M, Christensen JJ, Overgaard J. Morbidity and mortality of ischaemic heart disease in high-risk breast-cancer patients after adjuvant postmastectomy systemic treatment with or without radiotherapy: analysis of DBCG 82b and 82c randomised trials. Radiotherapy Committee of the Danish Breast Cancer Cooperative Group. Lancet. 1999 Oct 23;354(9188):1425-30. doi: 10.1016/s0140-6736(99)02245-x. PMID 10543669
- [Background] Emami B, Lyman J, Brown A, Coia L, Goitein M, Munzenrider JE, Shank B, Solin LJ, Wesson M. Tolerance of normal tissue to therapeutic irradiation. Int J Radiat Oncol Biol Phys. 1991 May 15;21(1):109-22. doi: 10.1016/0360-3016(91)90171-y. PMID 2032882
- [Background] Marks LB, Yu X, Prosnitz RG, Zhou SM, Hardenbergh PH, Blazing M, Hollis D, Lind P, Tisch A, Wong TZ, Borges-Neto S. The incidence and functional consequences of RT-associated cardiac perfusion defects. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):214-23. doi: 10.1016/j.ijrobp.2005.01.029. PMID 16111592
- [Background] Pierce SM, Recht A, Lingos TI, Abner A, Vicini F, Silver B, Herzog A, Harris JR. Long-term radiation complications following conservative surgery (CS) and radiation therapy (RT) in patients with early stage breast cancer. Int J Radiat Oncol Biol Phys. 1992;23(5):915-23. doi: 10.1016/0360-3016(92)90895-o. PMID 1639653
- [Background] Bradley J, Graham MV, Winter K, Purdy JA, Komaki R, Roa WH, Ryu JK, Bosch W, Emami B. Toxicity and outcome results of RTOG 9311: a phase I-II dose-escalation study using three-dimensional conformal radiotherapy in patients with inoperable non-small-cell lung carcinoma. Int J Radiat Oncol Biol Phys. 2005 Feb 1;61(2):318-28. doi: 10.1016/j.ijrobp.2004.06.260. PMID 15667949
- [Background] Pierce LJ. The use of radiotherapy after mastectomy: a review of the literature. J Clin Oncol. 2005 Mar 10;23(8):1706-17. doi: 10.1200/JCO.2005.08.109. No abstract available. PMID 15755979
- [Background] Campone M, Fumoleau P, Bourbouloux E, Kerbrat P, Roche H. Taxanes in adjuvant breast cancer setting: which standard in Europe? Crit Rev Oncol Hematol. 2005 Sep;55(3):167-75. doi: 10.1016/j.critrevonc.2005.04.003. PMID 16039867
- [Background] Giordano SH, Duan Z, Kuo YF, Hortobagyi GN, Freeman J, Goodwin JS. Impact of a scientific presentation on community treatment patterns for primary breast cancer. J Natl Cancer Inst. 2006 Mar 15;98(6):382-8. doi: 10.1093/jnci/djj090. PMID 16537830
- [Background] Taghian AG, Assaad SI, Niemierko A, Kuter I, Younger J, Schoenthaler R, Roche M, Powell SN. Risk of pneumonitis in breast cancer patients treated with radiation therapy and combination chemotherapy with paclitaxel. J Natl Cancer Inst. 2001 Dec 5;93(23):1806-11. doi: 10.1093/jnci/93.23.1806. PMID 11734597
- [Background] Burstein HJ, Bellon JR, Galper S, Lu HM, Kuter I, Taghian AG, Wong J, Gelman R, Bunnell CA, Parker LM, Garber JE, Winer EP, Harris JR, Powell SN. Prospective evaluation of concurrent paclitaxel and radiation therapy after adjuvant doxorubicin and cyclophosphamide chemotherapy for Stage II or III breast cancer. Int J Radiat Oncol Biol Phys. 2006 Feb 1;64(2):496-504. doi: 10.1016/j.ijrobp.2005.07.975. Epub 2005 Oct 21. PMID 16243442
- [Background] Voduc KD, Tyldesley S, Chia S. Risk of radiation pneumonitis in breast cancer patients treated with adjuvant taxanes and radiation. Vol 22; 2004. pp. 624-.
- [Background] Yu TK, Whitman GJ, Thames HD, Buzdar AU, Strom EA, Perkins GH, Schechter NR, McNeese MD, Kau SW, Thomas ES, Hortobagyi GN, Buchholz TA. Clinically relevant pneumonitis after sequential paclitaxel-based chemotherapy and radiotherapy in breast cancer patients. J Natl Cancer Inst. 2004 Nov 17;96(22):1676-81. doi: 10.1093/jnci/djh315. PMID 15547180
- [Background] Lind PA, Marks LB, Hardenbergh PH, Clough R, Fan M, Hollis D, Hernando ML, Lucas D, Piepgrass A, Prosnitz LR. Technical factors associated with radiation pneumonitis after local +/- regional radiation therapy for breast cancer. Int J Radiat Oncol Biol Phys. 2002 Jan 1;52(1):137-43. doi: 10.1016/s0360-3016(01)01715-1. PMID 11777631
- [Background] Beal K, Hudis C, Norton L, Wagman R, McCormick B. Radiation pneumonitis in breast cancer patients treated with taxanes: does sequential radiation therapy lower the risk? Breast J. 2005 Sep-Oct;11(5):317-20. doi: 10.1111/j.1075-122X.2005.21696.x. PMID 16174151
- [Background] Jaen J, Vazquez G, Alonso E, Leon A, Guerrero R, Almansa JF. Changes in pulmonary function after incidental lung irradiation for breast cancer: A prospective study. Int J Radiat Oncol Biol Phys. 2006 Aug 1;65(5):1381-8. doi: 10.1016/j.ijrobp.2006.03.008. Epub 2006 Jun 6. PMID 16757130
- [Background] Fan M, Marks LB, Lind P, Hollis D, Woel RT, Bentel GG, Anscher MS, Shafman TD, Coleman RE, Jaszczak RJ, Munley MT. Relating radiation-induced regional lung injury to changes in pulmonary function tests. Int J Radiat Oncol Biol Phys. 2001 Oct 1;51(2):311-7. doi: 10.1016/s0360-3016(01)01619-4. PMID 11567804
- [Background] Lind PA, Marks LB, Jamieson TA, Carter DL, Vredenburgh JJ, Folz RJ, Prosnitz LR. Predictors for pneumonitis during locoregional radiotherapy in high-risk patients with breast carcinoma treated with high-dose chemotherapy and stem-cell rescue. Cancer. 2002 Jun 1;94(11):2821-9. doi: 10.1002/cncr.10573. PMID 12115368
- [Background] Aitken RJ, Gaze MN, Rodger A, Chetty U, Forrest AP. Arm morbidity within a trial of mastectomy and either nodal sample with selective radiotherapy or axillary clearance. Br J Surg. 1989 Jun;76(6):568-71. doi: 10.1002/bjs.1800760613. PMID 2758260
- [Background] Bentzen SM, Dische S. Morbidity related to axillary irradiation in the treatment of breast cancer. Acta Oncol. 2000;39(3):337-47. doi: 10.1080/028418600750013113. PMID 10987231
- [Background] Bentzen SM, Overgaard M, Thames HD. Fractionation sensitivity of a functional endpoint: impaired shoulder movement after post-mastectomy radiotherapy. Int J Radiat Oncol Biol Phys. 1989 Sep;17(3):531-7. doi: 10.1016/0360-3016(89)90103-x. PMID 2506157
- [Background] Fathers E, Thrush D, Huson SM, Norman A. Radiation-induced brachial plexopathy in women treated for carcinoma of the breast. Clin Rehabil. 2002 Mar;16(2):160-5. doi: 10.1191/0269215502cr470oa. PMID 11911514
- [Background] Gerard JM, Franck N, Moussa Z, Hildebrand J. Acute ischemic brachial plexus neuropathy following radiation therapy. Neurology. 1989 Mar;39(3):450-1. doi: 10.1212/wnl.39.3.450. No abstract available. PMID 2927663
- [Background] Gerber L, Lampert M, Wood C, Duncan M, D'Angelo T, Schain W, McDonald H, Danforth D, Findlay P, Glatstein E, et al. Comparison of pain, motion, and edema after modified radical mastectomy vs. local excision with axillary dissection and radiation. Breast Cancer Res Treat. 1992;21(2):139-45. doi: 10.1007/BF01836960. PMID 1627817
- [Background] Lotze MT, Duncan MA, Gerber LH, Woltering EA, Rosenberg SA. Early versus delayed shoulder motion following axillary dissection: a randomized prospective study. Ann Surg. 1981 Mar;193(3):288-95. doi: 10.1097/00000658-198103000-00007. PMID 7011221
- [Background] Gillette EL, Mahler PA, Powers BE, Gillette SM, Vujaskovic Z. Late radiation injury to muscle and peripheral nerves. Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1309-18. doi: 10.1016/0360-3016(94)00422-H. PMID 7713790
- [Background] Haid A, Kuehn T, Konstantiniuk P, Koberle-Wuhrer R, Knauer M, Kreienberg R, Zimmermann G. Shoulder-arm morbidity following axillary dissection and sentinel node only biopsy for breast cancer. Eur J Surg Oncol. 2002 Nov;28(7):705-10. doi: 10.1053/ejso.2002.1327. PMID 12431466
- [Background] Harper CM Jr, Thomas JE, Cascino TL, Litchy WJ. Distinction between neoplastic and radiation-induced brachial plexopathy, with emphasis on the role of EMG. Neurology. 1989 Apr;39(4):502-6. doi: 10.1212/wnl.39.4.502. PMID 2538777
- [Background] Johansson S, Svensson H, Denekamp J. Dose response and latency for radiation-induced fibrosis, edema, and neuropathy in breast cancer patients. Int J Radiat Oncol Biol Phys. 2002 Apr 1;52(5):1207-19. doi: 10.1016/s0360-3016(01)02743-2. PMID 11955731
- [Background] Johansson S, Svensson H, Denekamp J. Timescale of evolution of late radiation injury after postoperative radiotherapy of breast cancer patients. Int J Radiat Oncol Biol Phys. 2000 Oct 1;48(3):745-50. doi: 10.1016/s0360-3016(00)00674-x. PMID 11020571
- [Background] Johansson S, Svensson H, Larsson LG, Denekamp J. Brachial plexopathy after postoperative radiotherapy of breast cancer patients--a long-term follow-up. Acta Oncol. 2000;39(3):373-82. doi: 10.1080/028418600750013140. PMID 10987234
- [Background] Keramopoulos A, Tsionou C, Minaretzis D, Michalas S, Aravantinos D. Arm morbidity following treatment of breast cancer with total axillary dissection: a multivariated approach. Oncology. 1993 Nov-Dec;50(6):445-9. doi: 10.1159/000227227. PMID 8233285
- [Background] Olsen NK, Pfeiffer P, Mondrup K, Rose C. Radiation-induced brachial plexus neuropathy in breast cancer patients. Acta Oncol. 1990;29(7):885-90. doi: 10.3109/02841869009096384. PMID 2261203
- [Background] Ryttov N, Holm NV, Qvist N, Blichert-Toft M. Influence of adjuvant irradiation on the development of late arm lymphedema and impaired shoulder mobility after mastectomy for carcinoma of the breast. Acta Oncol. 1988;27(6A):667-70. doi: 10.3109/02841868809091766. PMID 3219220
- [Background] Stoll BA, Andrews JT. Radiation-induced Peripheral Neuropathy. Br Med J. 1966 Apr 2;1(5491):834-7. doi: 10.1136/bmj.1.5491.834. No abstract available. PMID 20790877
- [Background] Swedborg I, Wallgren A. The effect of pre- and postmastectomy radiotherapy on the degree of edema, shoulder-joint mobility, and gripping force. Cancer. 1981 Mar 1;47(5):877-81. doi: 10.1002/1097-0142(19810301)47:53.0.co;2-3. PMID 7013962
- [Background] Tengrup I, Tennvall-Nittby L, Christiansson I, Laurin M. Arm morbidity after breast-conserving therapy for breast cancer. Acta Oncol. 2000;39(3):393-7. doi: 10.1080/028418600750013177. PMID 10987237
- [Background] Thompson AM, Air M, Jack WJL, et al. Arm morbidity after breast conservation and axillary therapy. The Breast 1995;4:273-276.
- [Background] Hack TF, Cohen L, Katz J, Robson LS, Goss P. Physical and psychological morbidity after axillary lymph node dissection for breast cancer. J Clin Oncol. 1999 Jan;17(1):143-9. doi: 10.1200/JCO.1999.17.1.143. PMID 10458227
- [Background] Warmuth MA, Bowen G, Prosnitz LR, Chu L, Broadwater G, Peterson B, Leight G, Winer EP. Complications of axillary lymph node dissection for carcinoma of the breast: a report based on a patient survey. Cancer. 1998 Oct 1;83(7):1362-8. doi: 10.1002/(sici)1097-0142(19981001)83:73.0.co;2-2. PMID 9762937
- [Background] Blomqvist L, Stark B, Engler N, Malm M. Evaluation of arm and shoulder mobility and strength after modified radical mastectomy and radiotherapy. Acta Oncol. 2004;43(3):280-3. doi: 10.1080/02841860410026170. PMID 15244252
- [Background] Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704. doi: 10.2106/JBJS.E.00835. PMID 16882890
- [Background] Middleton WD, Teefey SA, Yamaguchi K. Sonography of the rotator cuff: analysis of interobserver variability. AJR Am J Roentgenol. 2004 Nov;183(5):1465-8. doi: 10.2214/ajr.183.5.1831465. PMID 15505321
- [Background] Teefey SA, Rubin DA, Middleton WD, Hildebolt CF, Leibold RA, Yamaguchi K. Detection and quantification of rotator cuff tears. Comparison of ultrasonographic, magnetic resonance imaging, and arthroscopic findings in seventy-one consecutive cases. J Bone Joint Surg Am. 2004 Apr;86(4):708-16. PMID 15069134
- [Background] Kori SH, Foley KM, Posner JB. Brachial plexus lesions in patients with cancer: 100 cases. Neurology. 1981 Jan;31(1):45-50. doi: 10.1212/wnl.31.1.45. PMID 6256684
- [Background] Mondrup K, Olsen NK, Pfeiffer P, Rose C. Clinical and electrodiagnostic findings in breast cancer patients with radiation-induced brachial plexus neuropathy. Acta Neurol Scand. 1990 Feb;81(2):153-8. doi: 10.1111/j.1600-0404.1990.tb00952.x. PMID 2327236
- [Background] Moskovitz AH, Anderson BO, Yeung RS, Byrd DR, Lawton TJ, Moe RE. Axillary web syndrome after axillary dissection. Am J Surg. 2001 May;181(5):434-9. doi: 10.1016/s0002-9610(01)00602-x. PMID 11448437
- [Background] Leidenius M, Leppanen E, Krogerus L, von Smitten K. Motion restriction and axillary web syndrome after sentinel node biopsy and axillary clearance in breast cancer. Am J Surg. 2003 Feb;185(2):127-30. doi: 10.1016/s0002-9610(02)01214-x. PMID 12559441
- [Background] Maunsell E, Brisson J, Deschenes L. Arm problems and psychological distress after surgery for breast cancer. Can J Surg. 1993 Aug;36(4):315-20. PMID 8370012
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Hunsaker FG, Cioffi DA, Amadio PC, Wright JG, Caughlin B. The American academy of orthopaedic surgeons outcomes instruments: normative values from the general population. J Bone Joint Surg Am. 2002 Feb;84(2):208-15. doi: 10.2106/00004623-200202000-00007. PMID 11861726
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fayers P AN, Bjordal K, Groenvold M, Curran D, Bottomley A, on behalf of the EORTC Quality of Life Study Group. The EORTC QLQ-C30 Scoring Manual (3rd Edition). Brussels: European Organization for Research and Treatment of Cancer; 2001.
- [Background] Groenvold M, Klee MC, Sprangers MA, Aaronson NK. Validation of the EORTC QLQ-C30 quality of life questionnaire through combined qualitative and quantitative assessment of patient-observer agreement. J Clin Epidemiol. 1997 Apr;50(4):441-50. doi: 10.1016/s0895-4356(96)00428-3. PMID 9179103
- [Background] McLachlan SA, Devins GM, Goodwin PJ. Validation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) as a measure of psychosocial function in breast cancer patients. Eur J Cancer. 1998 Mar;34(4):510-7. doi: 10.1016/s0959-8049(97)10076-4. PMID 9713301
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Krueger EA, Fraass BA, McShan DL, Marsh R, Pierce LJ. Potential gains for irradiation of chest wall and regional nodes with intensity modulated radiotherapy. Int J Radiat Oncol Biol Phys. 2003 Jul 15;56(4):1023-37. doi: 10.1016/s0360-3016(03)00183-4. PMID 12829138
- [Background] Cho BC, Hurkmans CW, Damen EM, Zijp LJ, Mijnheer BJ. Intensity modulated versus non-intensity modulated radiotherapy in the treatment of the left breast and upper internal mammary lymph node chain: a comparative planning study. Radiother Oncol. 2002 Feb;62(2):127-36. doi: 10.1016/s0167-8140(01)00472-8. PMID 11937239
- [Background] Welsh JS, Patel RR, Ritter MA, Harari PM, Mackie TR, Mehta MP. Helical tomotherapy: an innovative technology and approach to radiation therapy. Technol Cancer Res Treat. 2002 Aug;1(4):311-6. doi: 10.1177/153303460200100413. PMID 12625791
- [Background] Ruchala KJ, Olivera GH, Kapatoes JM, Schloesser EA, Reckwerdt PJ, Mackie TR. Megavoltage CT image reconstruction during tomotherapy treatments. Phys Med Biol. 2000 Dec;45(12):3545-62. doi: 10.1088/0031-9155/45/12/303. PMID 11131183
- [Background] Ding GX, Duggan DM, Coffey CW. Characteristics of kilovoltage x-ray beams used for cone-beam computed tomography in radiation therapy. Phys Med Biol. 2007 Mar 21;52(6):1595-615. doi: 10.1088/0031-9155/52/6/004. Epub 2007 Feb 27. PMID 17327651
- [Background] Huntzinger C, Munro P, Johnson S, Miettinen M, Zankowski C, Ahlstrom G, Glettig R, Filliberti R, Kaissl W, Kamber M, Amstutz M, Bouchet L, Klebanov D, Mostafavi H, Stark R. Dynamic targeting image-guided radiotherapy. Med Dosim. 2006 Summer;31(2):113-25. doi: 10.1016/j.meddos.2005.12.014. PMID 16690452
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu